CLINICAL TRIAL: NCT04807309
Title: PRETELL: PREvention of TELomere-related Complications After Lung Transplant
Acronym: PRETELL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Souheil El-Chemaly, MD, MPH, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021P000271
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Short Telomere Length; Lung Transplant
Keywords: Danazol; Short telomere; Lung transplant; Prevention; Leukopenia
MeSH Terms: conditions — Leukopenia | interventions — Danazol

STUDY DESIGN:
Intervention Model Description: Randomized double blind 2:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Similar tablets will be generated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo comparison
  Interventions: Drug: Placebo
- Danazol Pill (Active Comparator): Danazol 200mg orally twice a day
  Interventions: Drug: Danazol Pill

INTERVENTIONS:
Drug: Danazol Pill — Danazol 200 mg orally twice a day
  Arms: Danazol Pill
Drug: Placebo — Placebo twice a day
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of Danzol in lung transplant recipients with short telomeres.

Subjects with short telomeres recipient of lung transplant, will be randomized in the first month post-transplant to either placebo or Danazol (200mg bid) in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. Ability to give informed consent
3. Recipient of lung transplantation
4. Short telomeres assessed either pre-transplant or post-transplant with FLOW-FISH as lymphocyte telomere length <10th percentile predicted for age
5. Clinically stable one month after lung transplant

Exclusion Criteria:

1. Patients on androgen hormones to include testosterone or high dose estrogen (estradiol 0.5 mg/day or greater) during 12 months prior to enrollment
2. Patients with active thrombosis or thromboembolic disease and history of such events unless thrombosis is line related.
3. Undiagnosed abnormal genital bleeding, porphyria, androgen-dependent tumor, or prostatic hypertrophy
4. Patients with active hepatitis B or C
5. Patients who have received a bone marrow transplant
6. Clinically unstable after lung transplantation
7. Current pregnancy, or unwillingness to take be on two forms of contraceptives including a barrier method of birth control or practice abstinence to refrain from pregnancy if of childbearing potential during the course of the study
8. Lactating women, due to the potentially harmful effects on the nursing child
9. Patients with abnormal liver function AST, ALT >3 times normal
10. Subjects with a history of benign intracranial hypertension
11. Subjects with a history of liver disease not limited to alcoholic hepatitis/cirrhosis, non-alcoholic steatohepatitis (NASH), autoimmune hepatitis (AIH), primary biliary cirrhosis (PBC), and/or history of hepatic adenoma.
12. Subjects with poorly controlled or uncontrolled Type I or II diabetes mellitus
13. Significant renal abnormalities GFR< 40 ml/min/m2
14. Significant cardiac dysfunction with ejection fraction less than 50%
15. Moribund status such as death is expected in the coming year
16. Currently taking carbamazepine, pimozide or lomitapide
17. Inability to understand the investigational nature of the study or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 weeks
  The incidence, severity, outcome, and relationship to study treatment of adverse events and serious adverse events.
  Change from baseline in clinical laboratory test results.

SECONDARY OUTCOMES:
Occurrence of WBC <2000/µl | 48 weeks
  -Occurrence of WBC <2000/µl at any time during study period.
Cumulative number of events where WBC < 2000/µl | 48 weeks
  - Evaluating cumulative number of events where WBC < 2000/µl

OTHER OUTCOMES:
Telomere length | 48 weeks
  -Measure change in lymphocyte telomere length at end of study drug administration compared to screening

IPD SHARING:
Plan to Share IPD: No